CLINICAL TRIAL: NCT03114683
Title: Efficacy and Safety Evaluation of IBI308 in Treatment of Patients With Relapsed/Refractory Classical Hodgkin's Lymphoma: a Multicenter, Single Arm, Phase II Study
Brief Title: Efficacy and Safety Evaluation of IBI308 in Treatment of Patients With Relapsed/Refractory Classical Hodgkin's Lymphoma
Acronym: ORIENT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308B201
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Relapsed/Refractory Classical Hodgkin's Lymphoma
Keywords: Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI308 (Experimental)
  Interventions: Drug: PD1

INTERVENTIONS:
Drug: PD1 — IBI308 200mg/3 weeks

SUMMARY:
The study is to evaluate ORR, CR, PR DCR DOR PFS and safety of IBI308 in treatment of patients with Relapsed/Refractory Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Patients with classical Hodgkin lymphoma(cHL) who relapse after autologous stem-cell transplantation(ASCT) or progress after multiple lines of chemotherapy have a poor prognosis, with a median survival of approximately 1.2 years.

CHL frequently harbors a spectrum of chromosome 9p24.1/PD-L1/PD-L2 alterations, leading to overexpression of the programmed death 1 ligands,PD-L1 and PD-L2.

Sintilimab is a humanized monoclonal antibody against PD-1 that blocks the interaction between PD-1 and its ligands and was approved for relapsed/refractory Hodgkin lymphoma in China in 2018.

This study is a single arm,phase 2 study designed to evaluate the clinical activity of sintilimab in Chinese patients with R/R

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological confirmed classical Hodgkin's lymphoma (cHL).
2. Relapsed/refractory cHL, which failed second line and above therapy (including radiotherapy and autologous hematopoietic stem cell transplantation, ASCT); subject with no response to or with progression after ASCT is eligible.
3. At least one measurable disease (long axis>15 mm or short axis>10 mm, with uptake on 18FDG-PET)
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2.
5. Signed written informed consent form and willing and able to comply with scheduled visits and other requirements of the study.
6. Age ≥ 18.
7. Life expectancy of at least 12 weeks.
8. Subjects of reproductive potential must be willing to use adequate contraception during the course of the study and through 90 days after the last dose of study medication.
9. Adequate organ and bone marrow function:

   1. Count of Blood Cells: absolute neutrophil count (ANC) ≥ 0.75 × 109 / L; platelet count (PLT) ≥ 50 × 109 / L; hemoglobin content (HGB) ≥ 8.0 g / dL; no granulocyte colony-stimulating factor, platelet or red blood cells infusion in the last 14 days.
   2. Liver function: total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
   3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN.
   4. Thyroid function: thyroid stimulating hormone (TSH) in normal range (TSH abnormalities due to non-autoimmune causes can be enrolled).

Exclusion Criteria:

1. Known nodular lymphocyte predominant Hodgkin lymphoma.
2. Known central nervous system lymphoma.
3. Received ASCT within 90 days of the first dose of study medication.
4. Prior exposure to any anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody.
5. Currently participating in an interventional clinical study, unless participating in observational study or during follow-up period of an interventional study.
6. Received any investigational agent within 4 weeks of the first dose of study medication.
7. Received last dose of radiotherapy or anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy or arterial embolization) within 3 weeks of the first dose of study medication; received last dose of nitrosourea or mitomycin C within 6 weeks of the first dose of study medication.
8. Received systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks of first dose. Inhaled or topical steroids and adrenal replacement steroid doses are permitted in the absence of active autoimmune disease.
9. Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
10. Underwent major operation (craniotomy, thoracotomy or laparotomy) within 4 weeks of the first dose of study medication or open wound, ulcer or fracture.
11. Activated, known or suspected autoimmune diseases or history of the disease with two years before enrollment. Vitiligo, psoriasis, hair loss, or Graves disease which do not need systemic treatment in 2 years, or hypothyroidism which only need thyroid hormone replacement therapy, or type-1 diabetes which only need insulin replacement therapy is eligible for enrollment.
12. Known primary immunodeficiency disorders.
13. Active tuberculosis.
14. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation.
15. Known allergy or hypersensitivity to any monoclonal antibodies or any components used in their preparation.
16. Uncontrolled concomitant disease, including but not limited to :

    1. Human Immunodeficiency Virus (HIV) infection (HIV antibody positive)
    2. Active or poorly controlled severe infection
    3. Symptomatic congestive heart failure (New York Heart Association grade Ⅲ-IV) or symptomatic, poorly controlled arrhythmia
    4. Poorly controlled arterial hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg) with standard treatment
    5. Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke or transient ischemic attack, within 6 months before enrollment
    6. Prior life-threatening blood loss or grade 3/4 gastrointestinal/varicosity bleeding requiring blood infusion, endoscopic or surgical intervention within 3 months of enrollment
    7. Prior deep vein thrombosis, pulmonary embolism or any other severe thromboembolism events (implanted port or catheter caused thrombosis, or superficial vein thrombosis are not considered as severe thromboembolism events) within 3 months before enrollment
    8. History of uncontrolled metabolic disorder, non-malignant organ or systemic disease or secondary carcinomatous reaction, with high medical risk and/or uncertainty of survival evaluation
    9. With hepatic encephalopathy, hepato-renal syndrome or hepatic cirrhosis of Child-Pugh grade B or higher.
    10. History of intestinal obstruction or the following diseases: inflammatory bowel disease or extensive bowel resection (partial colonic resection or extensive small bowel resection, concomitant with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea
    11. Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study
17. Known acute or chronic active hepatitis B infection (chronic HBV carrier or non-active HBsAg positive subject is eligible) or acute or chronic active hepatitis C (HCV antibody negative subject is eligible; HCV RNA examination is required for HCV antibody positive subject, subject is eligible for enrollment if result was negative)
18. History of gastrointestinal perforation and /or fistula within 6 months before enrollment
19. Subjects with interstitial lung disease
20. Uncontrolled third space effusion, e.g. ascites or pleural effusion cannot be drained or controlled
21. Other primary malignancy, with the exception of:

    1. Curable malignancy (e.g. papillary thyroid carcinoma)
    2. Without active disease in the last 5 years and with very low recurrence risk
    3. Non-melanoma skin cancer or malignant freckle-like nevus with adequate treatment and no evidence of recurrence ;
    4. Adequately treated in-situ carcinoma
22. Women who are pregnant or in lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Chinese academy of Medical sciences, Beijing, China

REFERENCES:
- [Background] Shi Y, Su H, Song Y, Jiang W, Sun X, Qian W, Zhang W, Gao Y, Jin Z, Zhou J, Jin C, Zou L, Qiu L, Li W, Yang J, Hou M, Zeng S, Zhang Q, Hu J, Zhou H, Xiong Y, Liu P. Safety and activity of sintilimab in patients with relapsed or refractory classical Hodgkin lymphoma (ORIENT-1): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2019 Jan;6(1):e12-e19. doi: 10.1016/S2352-3026(18)30192-3. PMID 30612710
- [Background] Shi Y, Su H, Song Y, Jiang W, Sun X, Qian W, Zhang W, Gao Y, Jin Z, Zhou J, Jin C, Zou L, Qiu L, Li W, Yang J, Hou M, Xiong Y, Zhou H, Du X, Wang X, Peng B. Circulating tumor DNA predicts response in Chinese patients with relapsed or refractory classical hodgkin lymphoma treated with sintilimab. EBioMedicine. 2020 Apr;54:102731. doi: 10.1016/j.ebiom.2020.102731. PMID 32304999
- See also: Lancet Haematology 2019;6:e12-19 — https://pubmed.ncbi.nlm.nih.gov/30612710/
- See also: Lancet Haematology 2019;6:e12-19 (full text) — https://pubmed.ncbi.nlm.nih.gov/32304999/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Update analysis data cutoff date of safety data: 30 Sep, 2019. Update analysis data cutoff date of efficacy data: 12 Feb, 2018.
Groups:
- Sintilimab: Subjects received sintilimab 200mg by intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 2 years
Period: Overall Study
Arm/Group | Sintilimab
Started | 96
Completed | 52
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Sintilimab
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.83 (10.884)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 96
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 96

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed According to the Revised International Working Group Response Criteria for Malignant Lymphoma in 2007(IWG 2007) by the Independent Radiological Review Committee (IRRC).
Description: Per Revised International Working Group Response Criteria for Malignant Lymphoma in 2007(IWG 2007) assessed by CT and PET: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), ≥50% decrease in SPD of up to 6 largest dominant masses, no increase in size of other nodes; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sintilimab
Number analyzed (Participants) | 96
percentage of participants | 85.4 [76.7 to 91.8]

ADVERSE EVENTS:
Time Frame: Cutoff date of 30 Sep,2019 Serious AEs: Up to 90 days after last administration of investigation products Other AEs: Up to 90 days after last administration of investigation products
Description: All adverse events, including serious adverse events, will be collected since the consent form is signed until 90th day after last administration of investigation products, either observed by investigator or by the spontaneous reported by subjects.
Arm/Group | Sintilimab
All-Cause Mortality (participants affected / at risk) | 3/96
Serious Adverse Events (participants affected / at risk) | 24/96
Other Adverse Events (participants affected / at risk) | 96/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=96)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Death (General disorders) | 2
Chest pain (General disorders) | 1
Mass (General disorders) | 1
Pyrexia (General disorders) | 1
Autoimmune myocarditis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Thyroiditis (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Myocardial necrosis marker increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=96)
Blood thyroid stimulating hormone increased (Investigations) | 31
Alanine aminotransferase increased (Investigations) | 28
Lymphocyte count decreased (Investigations) | 26
Neutrophil count decreased (Investigations) | 20
Weight increased (Investigations) | 19
White blood cell count decreased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 18
Blood uric acid increased (Investigations) | 15
Gamma-glutamyltransferase increased (Investigations) | 15
Platelet count decreased (Investigations) | 15
Thyroxine free decreased (Investigations) | 15
Blood lactate dehydrogenase increased (Investigations) | 12
Blood glucose increased (Investigations) | 11
Blood urine present (Investigations) | 11
Lipase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 9
Weight decreased (Investigations) | 9
Bilirubin conjugated increased (Investigations) | 8
Neutrophil count increased (Investigations) | 8
Protein urine present (Investigations) | 8
Blood creatine phosphokinase increased (Investigations) | 7
White blood cell count increased (Investigations) | 7
White blood cells urine positive (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 6
C-reactive protein increased (Investigations) | 6
Electrocardiogram T wave abnormal (Investigations) | 6
Haemoglobin decreased (Investigations) | 6
Lymphocyte percentage decreased (Investigations) | 6
Blood albumin decreased (Investigations) | 5
Blood creatinine increased (Investigations) | 5
Haemoglobin increased (Investigations) | 5
Tri-iodothyronine decreased (Investigations) | 5
Tri-iodothyronine free increased (Investigations) | 5
Pyrexia (General disorders) | 52
Asthenia (General disorders) | 6
Chills (General disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 27
Urinary tract infection (Infections and infestations) | 14
Lung infection (Infections and infestations) | 7
Viral upper respiratory tract infection (Infections and infestations) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Hypothyroidism (Endocrine disorders) | 21
Hyperthyroidism (Endocrine disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 14
Sinus tachycardia (Cardiac disorders) | 6
Sinus bradycardia (Cardiac disorders) | 5
Proteinuria (Renal and urinary disorders) | 10
Insomnia (Psychiatric disorders) | 6
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03114683/Prot_SAP_000.pdf